CLINICAL TRIAL: NCT02800772
Title: Impact of Intraduodenal Acetic Acid Infusion on Pancreatic Duct Cannulation During Endoscopic Retrograde Cholangiopancreatography: a Double-blind, Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Digestive Endoscopy Center, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ERCP-01
Record Dates: First submitted 2016-06-11; First posted 2016-06-15 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Pancreatic Duct Cannulation During Endoscopic Retrograde Choledochopancreatography
Keywords: pancreatic duct; ERCP; acetic acid
MeSH Terms: interventions — Acetic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- acetic acid (Experimental): spray 50ml acetic acid to duodenal bulb
  Interventions: Dietary Supplement: acetic acid
- saline (Placebo Comparator): spray 50ml saline to duodenal bulb
  Interventions: Dietary Supplement: saline

INTERVENTIONS:
Dietary Supplement: acetic acid
  Arms: acetic acid
Dietary Supplement: saline
  Arms: saline

SUMMARY:
Intraduodenal acetic acid can stimulate secretion of water and bicarbonate from pancreatic ductal cells. In this study, acetic acid spraying to duodenal bulb was compared with saline solution for the facilitation of pancreatic duct cannulation in patients.The primary outcome was successful deep pancreatic duct cannulation. The secondary outcomes were the appearance of the major and minor papillary orifice, pancreatic juice flow from the papilla, time to achieve deep pancreatic duct cannulation, and fluoroscopy time for deep pancreatic duct cannulation in the acetic acid group versus saline group.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were(1)those with intact native papilla (2)who underwent endoscopic retrograde choledochopancreatography for pancreatic duct, (3)age≥18 years，≦80years,and (4)agreement to participate in the study.

Exclusion Criteria:

* Exclusion criteria were (1) a previous sphincterotomy, (2) previous attempted or unsuccessful endoscopic retrograde choledochopancreatography with papillary manipulation, (3) indwelling biliary or pancreatic stent(s), (4) active acute pancreatitis, (5) altered/postsurgical anatomy, (6) history of gastroparesis, and (7) endoscopic retrograde choledochopancreatography for sphincter of Oddi (SO) manometry.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
cannulation time for deep pancreatic duct cannulation | 2 days
fluoroscopy time for deep pancreatic duct cannulation | 2 days

SECONDARY OUTCOMES:
pancreatic juice flow from the major papilla | 2 days
appearance of the major papillary orifice | 2 days

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Fang J, Wang SL, Zhao SB, Hu LH, Yao J, Shen Z, Gu L, Xia T, Cai Q, Li ZS, Bai Y. Impact of intraduodenal acetic acid infusion on pancreatic duct cannulation during endoscopic retrograde cholangiopancreatography: A double-blind, randomized controlled trial. J Gastroenterol Hepatol. 2018 Oct;33(10):1804-1810. doi: 10.1111/jgh.14148. Epub 2018 May 4. PMID 29633339